CLINICAL TRIAL: NCT05377632
Title: Comparing the Modified Novel Trans-Retro Approach vs Conventional Retroperitoneal Approach in Robotic-Assisted Renal Surgery: An Open Label Randomized Controlled Trial
Brief Title: Comparing Two Different Approaches in Robotic-Assisted Renal Surgery
Acronym: PIONEER-OPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lukas J Hefermehl (Other)
Collaborators: Kantonsspital Baden (Other)
Responsible Party: Sponsor-Investigator, Lukas J Hefermehl, Principal Investigator, Kantonsspital Baden
Organization: Kantonsspital Baden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIONEER-OPTICS
Record Dates: First submitted 2022-05-03; First posted 2022-05-17 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Renal Tumor
Keywords: robotic surgery; renal tumor
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Licensed Practical Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hybrid-Group (Active Comparator): Laparoscopic and Robotic-assisted combined (partial) nephrectomy via the hybrid (trans-peritoneal and retroperitoneal) access route
  Interventions: Procedure: Robotic-assisted laparoscopic partial nephrectomy (LPN) or laparoscopic nephrectomy (LN)
- Retroperitoneal-Group (Active Comparator): Robotic-assisted laparoscopic (partial) nephrectomy via the retroperitoneal access route
  Interventions: Procedure: Robotic-assisted laparoscopic partial nephrectomy (LPN) or laparoscopic nephrectomy (LN)

INTERVENTIONS:
Procedure: Robotic-assisted laparoscopic partial nephrectomy (LPN) or laparoscopic nephrectomy (LN) — laparoscopic partial nephrectomy (LPN) or laparoscopic nephrectomy (LN) include bilateral tumors or tumors in a solitary kidney. Relative indications include familial renal cancer syndromes such as Von Hippel-Lindau, hereditary leiomyomatosis, or hereditary papillary renal cell carcinoma. Patients with chronic kidney disease are generally offered nephron sparing surgery for hope of future renal function preservation. This reasoning also applies to those patients with preexisting diseases that may threaten a solitary kidney such as uncontrolled diabetes and hypertension.

SUMMARY:
The purpose of this study is to determine if the novel TR approach is superior to the standard RP approach. The anticipated study outcome is a time saving of at least 30% from first skin incision to detection of the renal artery compared to the conventional RP approach, and also a better workspace perception by the operating surgeon.

DETAILED DESCRIPTION:
The trans abdominal approach (TA) for total and partial nephrectomy (PN) has been widely adopted due to the easy trocar placement and the good working space. The retroperitoneal approach (RP) has gained popularity because the renal artery is often found fast and the operation remains in an anatomically separated space, making it preferable, especially for patients who underwent abdominal surgery in the past. However, both approaches face difficulties. Trocar placement for RP can be challenging, and the working space often is limited, while TA is impaired in cases of dorsal tumors and dissection of the renal artery can be challenging due to the anatomic localization dorsally to the renal vein. Up until now, no direct systematically and prospective comparison of these two approaches was performed.

The overall objective of this trial is to assess if the novel TR approach is superior to the conventional RP approach in performing robotic assisted (partial) nephrectomy. To date, no systematic, prospective, randomised study has been conducted on this topic and described in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient with a renal tumor or non-functionally kidney that is a candidate for robotic assisted surgery (RAS) nephrectomy or partial nephrectomy (PN)
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Renal vein tumor thrombus
* Pregnancy or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
detection of the renal artery | During procedure/surgery
  Time from first skin incision to detection of the renal artery [Time in minutes]

SECONDARY OUTCOMES:
Operative time | During procedure/surgery
  The time from [Skin Incision] to [Skin Closure] in minutes as documented in OR-Management Information System
Robot docking time | During procedure/surgery
  The time from [Skin Incision] to [robot docking] in minutes as documented in OR-Spreadsheet.
Instrument insertion time | During procedure/surgery
  The time from [Skin Incision] to [insertion of the last instrument] in minutes as documented in OR-Spreadsheet
Off-console time | During procedure/surgery
  The time from [Skin Incision] to [start of first instrument movement by console surgeon] in minutes as documented in OR-Spreadsheet
Ischemia time | During procedure/surgery
  The time from [Placement of clamp on artery] to [Release of clamp] in minutes indicated by the console surgeon documented by the anesthesiologist
Surgical conversion to open surgery | During procedure/surgery
  Conversion from robotic to open surgery
Surgical conversion to radical nephrectomy | During procedure/surgery
  Conversion partial to radical nephrectomy
Intraoperative blood loss | During procedure/surgery
  Volume of blood loss during the surgical procedure in mL
Console surgeons perception of Trocar placement and working space | During procedure/surgery
  Assessment via The surgical rating score (Likert-scale, 1-5, higher scores mean a better outcome)
Side assistants perception of Trocar placement and working space | During procedure/surgery
  Assessment via The surgical rating score (Likert-scale, 1-5, higher scores mean a better outcome)
Pain assessment | During the hospital stay (up to day 7)
  Assessment of pain level via the Visual Analogue Scale (VAS, 1-10, higher scores mean more pain)
Pain Management | During the hospital stay (up to day 7)
  Documentation of pain management (according to the WHO Analgesic Ladder, 1-4, higher scores mean more intense pain treatment)
Kidney function via the estimated glomerular filtration rate (eGRF) | During the hospital stay (up to day 7)
  Data will be gathered from routine examination, not a mandatory assessment (Lab value read-outs from in the clinical Information System) [ml/min/1,73 m2]
Post operative complications | Day 30
  Any Clavien-Dindo I-V post-operative complication (standard classification for complication in surgery
Length of stay Length of stay | During the hospital stay (up to day 7)
  Time from surgery to discharge in days [d]
Procedure related readmissions | Day 30
  Readmission that can be linked to the (partial) nephrectomy, binary [Yes/No]
Procedure related reoperations | Day 30
  Re-operation that can be linked to the partial nephrectomy, binary [Yes/No]
Comprehensive Complication Index | Day 30
  Any complication that occurred within 30 days post surgery, Scale [from 0 (no complication) to 100 (death)]

CONTACTS AND LOCATIONS:
Overall Officials: Lukas J Hefermehl, MD, Principal Investigator — Kantonsspital Baden
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No
The data that will be recorded in this study will be available on reasonable request from the PI